CLINICAL TRIAL: NCT05000372
Title: 68Ga-grazytracer PET/CT of Tumor Responses to Immunotherapy in Subjects with Solid Tumor or Lymphoma
Brief Title: 68Ga-grazytracer PET/CT of Tumor Responses to Immunotherapy
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Peking University Cancer Hospital & Institute (Other)
Collaborators: Peking University Health Science Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: 2021KT86
Record Dates: First submitted 2021-07-27; First posted 2021-08-11 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: Cancer
Keywords: PET/CT; Immunotherapy; Immune checkpoint inhibition; Granzyme B; 68Ga labeling
MeSH Terms: conditions — Neoplasms; Lipodystrophy, Congenital Generalized

STUDY DESIGN:
Intervention Model Description: Single Group Assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Feasibility and safety of 68Ga-grazytracer (Experimental): The purpose of the study is to evaluate the safety and early predictive performance of 68Ga-grazytracer for immunotherapy.
  Interventions: Drug: 68Ga-grazytracer

INTERVENTIONS:
Drug: 68Ga-grazytracer — 68Ga-grazytracer PET/CT: after intravenous injection of 2.96-3.7 MBq/kg body weight of quality-controlled 68Ga-grazytracer, a Biograph mCT Flow 64 scanner or Total-body PET/CT uEXPLORER scanner will be applied, and the scan range will be from the top of the head to 1/3 of the upper thigh.

SUMMARY:
This is an open-label positron emission tomography/computed tomography (PET/CT) study to investigate the safety and clinical predictive value of 68Ga-grazytracer in subjects with solid tumor or lymphoma receiving immunotherapy.

DETAILED DESCRIPTION:
The investigators recently developed a granzyme B-specific radiotracer named 68Ga-grazytracer. This clinical trial aims to investigate whether granzyme B PET imaging using 68Ga-grazytracer could early identify tumor responses to immune checkpoint inhibitory therapy or CAR-T therapy in subjects with solid tumor and lymphoma. PET/CT imaging of 68Ga-grazytracer will be performed in subjects after immunotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Participants who were diagnosed with malignant tumors;
2. Patients who were scheduled to receive immunotherapy based on a decision made by a multidisciplinary team;
3. participants who had no prior immunotherapy;
4. participants who had no regional therapy within 3 months;
5. Participants aged ≥18 years.

Exclusion Criteria:

1. participants with a concurrent disease that would impede the treatment regimen;
2. Participants who were unable or unwilling to provide written informed consent.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2021-09-22 (Actual); Primary Completion 2024-05-25 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Incidence of 68Ga-grazytracer-emergent Adverse Events | 3 year
  Any adverse events following the administration of the radiotracer will be monitored.
Biodistribution of 68Ga-grazytracer | 3 year
  The distribution of 68Ga-grazytracer in tumors and healthy tissues will be examined through total-body dynamic PET/CT imaging.
Analyzing the in vivo granzyme B-specificity of 68Ga-grazytracer | 3 year
  The specificity of 68Ga-grazytracer will be validated by correlating the immunohistochemistry results of granzyme B in either surgical or biopsy tissue samples with the standardized uptake values (SUV) of 68Ga-grazytracer in the tumors.
Assessing the early predictive value of 68Ga-grazytracer for immunotherapy response | 3 year
  Participants will be categorized into groups with high or low 68Ga-grazytracer uptake in tumor lesions. The progression-free survival and treatment response, as assessed by RECIST 1.1 criteria, will be compared across these groups.

SECONDARY OUTCOMES:
Correlation analysis of 68Ga-grazytracer uptake and tumor immune phenotype | 3 year
  Participants' tumors will be classified as either "desert" or "non-desert" based on immunohistochemistry staining of CD8 from tumor samples. Subsequently, the relationship between 68Ga-grazytracer uptake and the tumors' immune phenotype will be compared.

CONTACTS AND LOCATIONS:
Overall Officials: Nan Li, M.D., Study Director — Peking University Cancer Hospital & Institute; Zhaofei Liu, Ph.D., Study Director — Peking University; Zhi Yang, Ph.D., Study Director — Peking University Cancer Hospital & Institute
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shen X, Zhou H, Zhou X, Liu Z, Meng X, Zhang L, Song Y, Guo R, Wang F, Li K, Li W, Yang Z, Liu Z, Li N. 68Ga-grazytracer PET for noninvasive assessment of response to immunotherapy in solid tumors and lymphomas: a phase 1/2 clinical trial. Nat Commun. 2024 Oct 10;15(1):8791. doi: 10.1038/s41467-024-53197-2. PMID 39389969
- [Derived] Zhou H, Wang Y, Xu H, Shen X, Zhang T, Zhou X, Zeng Y, Li K, Zhang L, Zhu H, Yang X, Li N, Yang Z, Liu Z. Noninvasive interrogation of CD8+ T cell effector function for monitoring early tumor responses to immunotherapy. J Clin Invest. 2022 Aug 15;132(16):e161065. doi: 10.1172/JCI161065. PMID 35788116